CLINICAL TRIAL: NCT00334997
Title: Early Stage Glottic Cancer: Endoscopic Excision or Radiotherapy [EaStER]
Brief Title: Endoscopic Surgery or Radiation Therapy in Treating Patients With Stage 0, Stage I, or Stage II Laryngeal Cancer of the Glottis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000478790; CRUK-BRD/05/024; EU-20611; CRUK-EASTER; ISRCTN17541410
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-03

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage 0 laryngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms | interventions — Endoscopy; Laser Therapy; Radiotherapy

INTERVENTIONS:
Procedure: endoscopic surgery
Procedure: laser surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Endoscopic surgery is a less invasive type of surgery for laryngeal cancer and may have fewer side effects and improve recovery. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether endoscopic surgery is more effective than radiation therapy in treating laryngeal cancer of the glottis.

PURPOSE: This randomized phase II trial is studying endoscopic surgery to see how well it works compared with radiation therapy in treating patients with stage 0, stage I, or stage II laryngeal cancer of the glottis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of conducting a large phase III randomized study in the future, comparing radiotherapy vs endoscopic excision in patients with stage 0-II laryngeal cancer of the glottis.
* Determine patient acceptability of the proposed trial design.
* Compare the effect of using dedicated head and neck research nurses vs general nurses on patient recruitment.
* Refine outcome measures, including voice analysis and quality of life.

OUTLINE: This is a randomized, controlled, multicenter, pilot study. Patients are stratified according to participating center and T stage (Tis or T1 vs T2a). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo endoscopic excision via CO_2 laser or cold steel.
* Arm II: Patients undergo radiotherapy once daily, 5 days a week, for 3-4 weeks. Patients undergo vocal analysis at baseline and at 6 months and 1 and 2 years after randomization.

Quality of life is assessed at baseline, at 1 year, and then annually for 5 years.

After completion of study treatment, patients are followed periodically for up to 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the glottic larynx, including tumors at the anterior commissure

  * Stage 0-II (Tis, T1, or T2a)
* No clinical or radiological sign of nodal involvement
* No evidence of distant metastases
* Airway anatomy suitable for endoscopic excision

PATIENT CHARACTERISTICS:

* Fit to receive radical treatment as either radiotherapy or endoscopic excision
* Life expectancy ≥ 2 years
* No other cancer in the past 10 years except basal cell carcinoma of the skin or adequately treated carcinoma in situ of the uterine cervix
* No vasculitic conditions adversely affecting radiotherapy
* No other co-existing medical condition that would limit life expectancy
* Not pregnant

PRIOR CONCURRENT THERAPY:

* No concurrent chemotherapy
* No concurrent palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Feasibility
Patient acceptability

SECONDARY OUTCOMES:
Voice analysis
Quality of life
Economic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Birchall, MD, Study Chair — Southmead Hospital
Locations (6):
- United Kingdom (6):
  - Southmead Hospital, Bristol, England
  - Aintree University Hospital, Liverpool, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Royal Infirmary - Castle, Glasgow, Scotland